CLINICAL TRIAL: NCT01984840
Title: Effectiveness and Cost-effectiveness of Telemedicine for Chronic Obstructive Pulmonary Disease: The Danish "TeleCare North" Pragmatic Cluster-randomized Trial.
Brief Title: Telemedicine for Patients Suffering From COPD (Danish Telecare North Trial)
Acronym: TCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Ole K Hejlesen, PhD, Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RN-TN-001
Record Dates: First submitted 2013-06-14; First posted 2013-11-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Active Comparator): A tablet (a Samsung GALAXY TAB 2 (10.1)) that holds information on handling COPD in general and software that automatically instructs the patient in handling COPD during exacerbations. The device can also collect and transmit relevant disease-specific data, which are indicative of their current state of health, via an attached Fingertip Pulse Oximeter (Nonin, Onyx II % SpO2), a Digital Blood Pressure Monitor (Model UA-767, plus BT-C) and a scale. The device can measure four vital signs, which are transferred wirelessly: blood pressure, pulse, blood oxygen saturation and weight. The tablet can be activated and give a sound, when it is time for taking measurements again.
  Interventions: Device: Telemedicine
- Usual care (No Intervention): In Denmark, usual practice for treating, monitoring and caring for patients with COPD are the responsibility of the patient's general practitioner (treatment and monitoring) and the municipalities (practical help and nursing care). COPD patients can make appointments with their general practitioner or practice nurse free of charge in order to get help in managing COPD. Community based care and practical help varies. As a rule community care comes at regular intervals based on a clinically based estimate of the patients' needs, but the personnel are not necessarily certified nurses and often not fully educated in COPD and definitely not on call

INTERVENTIONS:
Device: Telemedicine
  Arms: Telemedicine

SUMMARY:
There are two main aims in this study. The first objective is to evaluate whether a particular telehealth solution, in addition to standard treatment and care, lead to a significant decrease in the mortality and an increase in health related quality of life for patients suffering from COPD that may benefit from telehealth compared with only standard treatment and care. The second objective is to examine the additional costs of the telehealth solution and assess whether this solution is a cost-effective way to care for patients with COPD across patients and municipality districts.

It is hypothesized that telehealth care will increase patients quality adjusted life years at both the cluster and individual level compared to usual practice, since no difference in mortality and a higher health related quality of life is expected. Furthermore, it is hoped that there will be a 30% reduction in the number of admissions and readmissions to hospitals and a 30% reduction in the number of outpatient visits resulting in fewer costs for hospitals. However, it is uncertain as to whether these savings are offset by other costs such as more visits to general practitioners, community care or the implementation costs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed COPD by spirometry
* in treatment corresponding to GOLD-guidelines
* motivated for treatment of COPD
* COPD is the primary disease
* fixed residence and be affiliated to a general practitioner in North Denmark Region
* At least one of the following criteria should also be met: MRCm (modified) ≥ 2 or MRC ≥3, CAT ≥ 10, have had at least 2 exacerbations within the last 12 months

Exclusion Criteria:

* no phone line or GSM coverage
* unable to understand Danish sufficiently to complete study questionnaires
* have a cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1225 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 12 month follow-up
  SF-36
Incremental cost-effectiveness ratio (ICER) | 12 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark

REFERENCES:
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Witt Udsen F, Lilholt PH, Hejlesen OK, Ehlers LH. Subgroup analysis of telehealthcare for patients with chronic obstructive pulmonary disease: the cluster-randomized Danish Telecare North Trial. Clinicoecon Outcomes Res. 2017 Jul 7;9:391-401. doi: 10.2147/CEOR.S139064. eCollection 2017. PMID 28740411
- [Derived] Witt Udsen F, Lilholt PH, Hejlesen O, Ehlers L. Cost-effectiveness of telehealthcare to patients with chronic obstructive pulmonary disease: results from the Danish 'TeleCare North' cluster-randomised trial. BMJ Open. 2017 May 17;7(5):e014616. doi: 10.1136/bmjopen-2016-014616. PMID 28515193
- [Derived] Lilholt PH, Witt Udsen F, Ehlers L, Hejlesen OK. Telehealthcare for patients suffering from chronic obstructive pulmonary disease: effects on health-related quality of life: results from the Danish 'TeleCare North' cluster-randomised trial. BMJ Open. 2017 May 9;7(5):e014587. doi: 10.1136/bmjopen-2016-014587. PMID 28490555
- [Derived] Lilholt PH, Schaarup C, Hejlesen OK. An Iterative, Mixed Usability Approach Applied to the Telekit System from the Danish TeleCare North Trial. Int J Telemed Appl. 2016;2016:6351734. doi: 10.1155/2016/6351734. Epub 2016 Nov 16. PMID 27974888
- [Derived] Udsen FW, Lilholt PH, Hejlesen O, Ehlers LH. Effectiveness and cost-effectiveness of telehealthcare for chronic obstructive pulmonary disease: study protocol for a cluster randomized controlled trial. Trials. 2014 May 21;15:178. doi: 10.1186/1745-6215-15-178. PMID 24886225